CLINICAL TRIAL: NCT04343118
Title: Do Patients Benefit From Elective Implant Removal Following Plate Osteosynthesis of Clavicle Fractures - a Prospective Trial
Brief Title: Benefit of Surgical Hardware Removal Following Clavicle Fracture
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Chlodwig Kirchhoff, Clinical Professor, Technical University of Munich
Other Study IDs: 089_2019ME
Record Dates: First submitted 2020-04-01; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Clavicle Fracture
MeSH Terms: interventions — Hardware Removal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group Removal: All patient receiving surgical removal of plate osteosynthesis
  Interventions: Procedure: Hardware Removal

INTERVENTIONS:
Procedure: Hardware Removal — elective removal of plate osteosynthesis at the clavicle

SUMMARY:
Little is known about the beneficial aspects of elective implant removal following plate osteosynthesis of displaced clavicle fractures.

DETAILED DESCRIPTION:
Elective implant removal accounts for up to 30% of all orthopaedic surgeries. While there is general acceptance about the need of implant removal for obvious reasons, such as infections or implant failure, little is known about the beneficial aspects in cases of minor reasons. Therefore, we initiated this study to define patients' benefit of elective implant removal following plate osteosynthesis of displaced clavicle fractures.

Patients and Methods Prospective evaluation of patients was conducted before implant removal and 6 weeks postoperative. Subjective and objective criteria included patients' satisfaction, pain rating on a visual analog scale (VAS) and active range of motion (ROM) pre- and 6 weeks postoperative. Functional scoring included the SPADI, DASH score, the Constant Score and the Munich Shoulder Questionnaire (MSQ).

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* Radiologically consolidated clavicle fracture
* following ORIF using a superior anatomically preformed locking plate
* asking for elective implant removal
* written informed consent.

Exclusion Criteria:

* Pregnancy
* Under-aged
* Delinquent patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requesting implant removal
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Shoulder function | 6 Week post surgery
  Munich Shoulder Questionnaire allowing for calculation of Constant Score (0-100), Dash (0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Chlodwig Kirchhoff, MD, Principal Investigator — Klinikum rechts der Isar, TU München
Locations (1):
- Klinik und Poliklinik für Unfallchirurgie, Klinikum rechts der Isar, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wurm M, Beirer M, Zyskowski M, Volk C, Schwarz A, Biberthaler P, Kirchhoff C, Cronlein M. Does implant removal of superior clavicle plate osteosynthesis affect the functional outcome: a prospective trial. Arch Orthop Trauma Surg. 2022 Jan;142(1):139-144. doi: 10.1007/s00402-020-03669-z. Epub 2020 Nov 1. PMID 33130933